CLINICAL TRIAL: NCT03504371
Title: The Analgesic Efficacy of Erector Spinae Block in Comparison to Thoracic Epidural Anesthesia in Patients Having Transthoracic Oesophygeal Surgical Procedures
Brief Title: The Analgesic Efficacy of Erector Spinae Block in Comparison to Thoracic Epidural Anesthesia in Oesophageal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, Hoda Shokri, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R19
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2018-04

CONDITIONS: Analgesic Efficacy
Keywords: oesophageal surgeries-epidural-erector block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bilateral erector spinae block (Active Comparator): The patient placed in a lateral position and ultrasound transducer placed 3 cm lateral to the T7 spinous process. Three muscles will be identified: trapezius, rhomboid major, and erector spinae. 8-cm 22-gauge block needle will be inserted in a cephalad-to-caudad direction until the tip lay in the interfascial plane between rhomboid major and erector spinae muscles, as evidenced by visualization of local anesthetic spreading in a linear pattern between erector spinae and the bony shadows of the transverse processes. 20 mL of 0.25% bupivacaine will be injected then it will be repeated on the other side in the same way without changing the position of the patient to achieve sensory block T5-T10 .
  Interventions: Device: bilateral erector spinae block
- Thoracic epidural anesthesia (Sham Comparator): an epidural catheter placed at the T7-8 interspace after proper sterilization and positioning of the patient in the sitting position then standard technique of application will be applied, then a test dose consists of 3 ml of 1.5% preservative free lidocaine will be injected followed by 5-6 ml of bupivacaine 0.25%
  Interventions: Device: Thoracic epidural anesthesia

INTERVENTIONS:
Device: bilateral erector spinae block — The patient placed in a lateral position and transducer placed in a longitudinal orientation 3 cm lateral to the T7 spinous process. Three muscles will be identified superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. An 8-cm 22-gauge block needle will be inserted in a cephalad-to-caudad direction until the tip lay in the interfascial plane between rhomboid major and erector spinae muscles, as evidenced by visualization of local anesthetic spreading in a linear pattern between erector spinae and the bony acoustic shadows of the transverse processes. 20 mL of 0.25% bupivacaine will be injected then it will be repeated on the other side and preformed in the same way to achieve sensory block T5-T10 .
  Arms: bilateral erector spinae block
Device: Thoracic epidural anesthesia — patients will receive TEA where an epidural catheter will be placed at the T7-8 interspace after proper sterilization and positioning of the patient in the sitting position then standard technique of application will be applied, then a test dose consists of 3 ml of 1.5% preservative free lidocaine with 1:200,000 epinephrine will be injected followed by 5-6 ml of bupivacaine 0.25%.
  Arms: Thoracic epidural anesthesia

SUMMARY:
a total of 80 patients age of 36 years old to 65 years old, (ASA) physical status I and II undergoing oesophageal procedures.The patients will randomised using concealed envelope method into 2 groups, allocation of patients to either group will be done by clinician not involved in the study. There are 2 groups of patients: TEA combined with GA (TEA group) or bilateral erector spinae block combined with GA (erector group). . In TEA group, patients will receive TEA where an epidural catheter will be placed at the T7-8 interspace after proper sterilization and positioning of the patient in the sitting position then standard technique of application will be applied, then a test dose consists of 3 ml of 1.5% preservative free lidocaine with 1:200,000 epinephrine will be injected followed by 5-6 ml of bupivacaine 0.25%. Anaesthesia will be standardised In the TEA group, an additional 4-5mL epidural doses of bupivacaine 0.25% will be administered at 1 h intervals. In the second group, patients will receive bilateral ESP block which will be performed as follows. The patient will be placed in a lateral position ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the T7 spinous process. Three muscles will be identified superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. An 8-cm 22-gauge block needle will be inserted in a cephalad-to-caudad direction until the tip lay in the interfascial plane between rhomboid major and erector spinae muscles, as evidenced by visualization of local anesthetic spreading in a linear pattern between erector spinae and the bony acoustic shadows of the transverse processes. A total of 20 mL of 0.25% bupivacaine will be injected then it will be repeated on the other side and preformed in the same way without changing the position of the patient to achieve sensory block T5-T10 .

DETAILED DESCRIPTION:
The patients will randomised into 2 groups. There are 2 groups of patients: TEA combined with GA or bilateral erector spinae block combined with G. In TEA group, patients will receive TEA, an epidural catheter will be placed at the T7-8 interspace after positioning of the patient in the sitting position then standard technique of application will be applied, then a test dose consists of 3 ml of 1.5% preservative free lidocaine with 1:200,000 epinephrine will be injected followed by 5-6 ml of bupivacaine 0.25%. Anaesthesia will be standardised. A left-sided, double-lumen thoracostomy tube will be inserted and confirmed by bronchofiberoscopy. In the TEA group, an additional 4-5mL epidural doses of bupivacaine 0.25% will be administered at 1 h intervals. In the second group, patients will receive bilateral ESP block which will be performed as follows. The patient will be placed in a lateral position and a high-frequency linear ultrasound transducer (GE LOGIQe, Wauwatosa, Wisconsin) will be placed in a longitudinal orientation 3 cm lateral to the T7 spinous process. Three muscles will be identified superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. An 8-cm 22-gauge block needle (EchoStim; Benlan Inc, Oakville, Canada) will be inserted in a cephalad-to-caudad direction until the tip lay in the interfascial plane between rhomboid major and erector spinae muscles, as evidenced by visualization of local anesthetic spreading in a linear pattern between erector spinae and the bony acoustic shadows of the transverse processes. A total of 20 mL of 0.25% bupivacaine will be injected then it will be repeated on the other side and preformed in the same way without changing the position of the patient to achieve sensory block T5-T10 .

Hemodynamics as heart rate, arterial blood pressure, central venous pressure and oxygen saturation will be monitored intraoperatively. The heart rate and arterial blood pressure will be maintained within 20% of the preoperative values.

At the end of the procedure, in both groups, anesthesia will be discontinued and neuromuscular blockade will be antagonized with neostigmine, intravenous (0.05 mg/kg) and atropine intravenous (0.03 mg/kg) at appropriate doses.

The patients will be transported postoperatively to the intensive care unit. if VAS > 5 , Patient-controlled analgesia using elastomeric pump will be established with IV doses of morphine in the erector group (basal rate about 0.5mg/h to 1 mg/h and bolus dose of 2 mg , 300 mL maximum dose) and epidural analgesia in the TEA group (top up doses of about 4 ml of bupivacaine 0.125% + morphine 20 μg/mL, bolus doses 2 mL to 3 mL, 300 ml maximum dose). The patients will be monitored in the postanaesthesia care unit (PACU)

ELIGIBILITY:
Inclusion Criteria:

36-65 years old oesophageal procedures ASA I,II

-

Exclusion Criteria:

* cardiac dysfunction Renal or hepatic impairment patient refusal Immune disorders Allergy to local anesthetics neuromuscular disorders

Ages: 36 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 24 h
  minor complications (hypotension, vomiting, urinary retention and catheter related complications) and major complications (mortality).

SECONDARY OUTCOMES:
length of hospital stay | 15-17 days
  Recovery time from end of surgery till discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Effat, Study Chair — Ain Shams University
Locations (1):
- Ain Shams U, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol statistical analysis
Supporting Information: Study Protocol
Time Frame: 6 months